CLINICAL TRIAL: NCT07250529
Title: Comparison of Left Bundle Branch Pacing Versus Conventional Right Ventricular Pacing on AHRE Burden in Patients With Preserved Left Ventricular Ejection Fraction and High Ventricular Pacing Dependency (LBBP-AHRE Trial): A Randomized Study
Brief Title: Left Bundle Branch Pacing vs Right Ventricular Pacing on AHRE Burden in Patients With Preserved LVEF
Acronym: LBBP-AHRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Georgios Leventopoulos, Assistant Professor of Cardiology - Electrophysiology Patras University Hospital, Greece, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UHP-LBBP-AHRE-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF); Pacemaker Therapy; Atrioventricular Block; Preserved Ejection Fraction
Keywords: Left bundle branch pacing; Cardiac electrophysiology; Right ventricular pacing; AHRE burden; Preserved ejection fraction
MeSH Terms: conditions — Atrial Fibrillation; Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Conventional Right Ventricular Pacing (Active Comparator): Procedure: Standard right ventricular septal pacing
  Description: Implantation of a dual-chamber pacemaker with the ventricular lead placed in the RV septum.
  At follow-up, the ventricular pacing percentage and pacing configuration will be noted.
  Interventions: Device: Right Ventricular Pacing
- Arm 2: Left Bundle Branch Pacing (LBBP) (Active Comparator): Procedure: Left bundle branch pacing lead implantation
  Description: Implantation of a dual-chamber pacemaker with the ventricular lead placed at the left bundle branch area.
  Physiological pacing will be programmed into the devices and, at follow-up, the percentage of spontaneous pacing will be noted.
  Interventions: Device: Left Bundle Branch Pacing

INTERVENTIONS:
Device: Right Ventricular Pacing — Implantation of a dual-chamber pacemaker with the ventricular lead placed in the RV septum.
  At follow-up, the ventricular pacing percentage and pacing configuration will be noted.
  All devices used in this study are commercially available in the European Union and carry a valid CE mark.
  Arms: Arm 1: Conventional Right Ventricular Pacing
Device: Left Bundle Branch Pacing — Implantation of a dual-chamber pacemaker with the ventricular lead placed at the left bundle branch area.
  Physiological pacing will be programmed into the devices and, at follow-up, the percentage of spontaneous pacing will be noted.
  All devices used in this study are commercially available in the European Union and carry a valid CE mark.
  Arms: Arm 2: Left Bundle Branch Pacing (LBBP)

SUMMARY:
This prospective, randomized controlled trial aims to evaluate the effect of left bundle branch pacing (LBBP) compared with conventional right ventricular (RV) pacing on the burden of atrial high-rate episodes (AHREs) in patients with preserved left ventricular ejection fraction (LVEF) who are expected to require frequent ventricular pacing.

Atrial High-Rate Episodes (AHREs) are defined as episodes of atrial tachyarrhythmia that are automatically recorded by device diagnostics and detected by implanted cardiac devices. These episodes usually have an atrial rate ≥170-190 beats per minute and a duration ≥6 minutes. AHREs are linked to a higher risk of thromboembolic events and clinical atrial fibrillation (AF), and they may indicate subclinical AF or other atrial tachyarrhythmias.

Chronic RV pacing has been linked to mechanical and electrical dyssynchrony, which may encourage atrial remodeling and the development of AF. LBBP provides a more physiological ventricular activation and may reduce atrial arrhythmic burden.

Patients with LVEF >50% and atrioventricular (AV) conduction disorders requiring a dual-chamber pacemaker will be randomized to either conventional RV septal pacing or LBBP.

DETAILED DESCRIPTION:
This prospective, randomized trial compares left bundle branch pacing (LBBP) with conventional right ventricular (RV) pacing in patients with preserved left ventricular ejection fraction (LVEF ≥50%) who are expected to require frequent ventricular pacing. The primary goal is to evaluate the effect of LBBP versus RV pacing on atrial high-rate episode (AHRE) burden, detected by dual-chamber pacemakers. AHREs are device-recorded atrial tachyarrhythmias (atrial rate ≥170-190 bpm, duration ≥6 minutes) associated with increased risk of atrial fibrillation (AF) and thromboembolic events.

Eligible patients with AV conduction disorders and sinus rhythm will be randomized 1:1 to LBBP or RV septal pacing at pacemaker implantation. All devices used are commercially available in the European Union and carry a valid CE mark. Device interrogation will occur at 3, 6, and 12 months to record AHRE burden, pacing percentage, and occurrence of AF. Permanent AF will be defined per ESC Guidelines, based on physician-patient consensus, including a rate-control strategy when rhythm restoration is not attempted.

Secondary outcomes include AHRE episode duration, progression to clinical AF, development of permanent AF, device- or procedure-related complications, hospitalization due to AF, need for cardioversion, and all-cause mortality. Beta-blocker therapy for other indications is allowed and documented.

This study will provide prospective, randomized evidence on whether physiological ventricular activation with LBBP reduces AHRE burden compared with conventional RV pacing in patients with preserved systolic function and high expected ventricular pacing dependency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled implantation of a dual-chamber pacemaker for:

Permanent complete heart block Permanent second-degree AV block (Mobitz II or Mobitz I)

* Documented preserved LVEF (≥50%)
* Sinus rhythm at baseline
* Ability to provide written informed consent

Exclusion Criteria:

* History of paroxysmal, persistent, or permanent atrial fibrillation
* Previous atrial fibrillation ablation (catheter-based or surgical)
* LVEF < 50%
* Sinus node disease
* Transient AV block requiring pacemaker implantation
* Significant structural or valvular heart disease
* Requirement for pacemaker system upgrade during the study period
* Requirement for antiarrhythmic therapy for causes other than atrial fibrillation
* Existing pacemaker or other cardiac device requiring modification for study participation
* Enrollment in another clinical trial that could interfere with study endpoints or pacing parameters
* Contraindication to LBBP or associated lead implantation procedure
* Life expectancy < 12 months
* Any condition judged by the investigator to compromise participation or the integrity of study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-11-25 (Estimated); Study Completion 2028-04-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of time in AHRE during the total monitored period (device-detected). | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
  Cumulative duration of all AHREs (>6 minutes) divided by total monitoring time, expressed as a percentage (aligning with current device-based burden metrics).

SECONDARY OUTCOMES:
Percentage of time in AHRE episodes of 6 minutes to 24 hours, expressed as a percentage of total monitored time. | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
Percentage of time in AHRE episodes >24 hours, expressed as a percentage of total monitored time. | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
Incidence of progression to clinically documented atrial fibrillation (paroxysmal or persistent, symptomatic or asymptomatic, confirmed by ECG, Holter, or wearable monitoring). | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
Development of permanent atrial fibrillation. | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
  Atrial fibrillation (AF) will be evaluated using routine interrogation of implanted pacemakers, which provide device-recorded atrial arrhythmia data, including AF burden and episode duration. Permanent atrial fibrillation will be defined according to the ESC Guidelines for Atrial Fibrillation and will require a consensus decision between the treating physician and the patient that the arrhythmia is ongoing. This consensus will also include an agreement to pursue a rate-control strategy with no further attempts to restore or maintain sinus rhythm.
Device- or procedure-related complications (e.g., cardiac perforation, pericardial tamponade, pneumothorax, hemothorax, infection requiring antibiotics or system removal, generator or lead malfunction, hematoma). | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
All-cause mortality. | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation
Hospitalization due to AF | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.
Need for cardioversion. | From pacemaker implantation (or randomization) to 12 months. All participants will be evaluated at 3, 6, and 12 months after pacemaker implantation.

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital of Patras, Pátrai, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Becher N, Metzner A, Toennis T, Kirchhof P, Schnabel RB. Atrial fibrillation burden: a new outcome predictor and therapeutic target. Eur Heart J. 2024 Aug 16;45(31):2824-2838. doi: 10.1093/eurheartj/ehae373. PMID 38953776
- [Result] Jansson V, Bergfeldt L, Schwieler J, Kenneback G, Rubulis A, Jensen SM, Raatikainen P, Sciaraffia E, Blomstrom-Lundqvist C. Atrial fibrillation burden, episode duration and frequency in relation to quality of life in patients with implantable cardiac monitor. Int J Cardiol Heart Vasc. 2021 May 11;34:100791. doi: 10.1016/j.ijcha.2021.100791. eCollection 2021 Jun. PMID 34036145
- [Result] Rosner GF, Reiffel JA, Hickey K. The Concept of "Burden" in Atrial Fibrillation. J Atr Fibrillation. 2012 Feb 2;4(5):400. doi: 10.4022/jafib.400. eCollection 2012 Feb-Mar. PMID 28496712
- [Result] Boriani G, Tartaglia E, Trapanese P, Tritto F, Gerra L, Bonini N, Vitolo M, Imberti JF, Mei DA. Subclinical atrial fibrillation/atrial high-rate episodes: what significance and decision-making? Eur Heart J Suppl. 2025 Feb 19;27(Suppl 1):i162-i166. doi: 10.1093/eurheartjsupp/suae088. eCollection 2025 Feb. PMID 39980773
- [Result] Simu G, Rosu R, Cismaru G, Puiu M, Gusetu G, Minciuna I, Istratoaie S, Tomoaia R, Zdrenghea D, Pop D. Atrial high-rate episodes: a comprehensive review. Cardiovasc J Afr. 2021 Mar-Apr 23;32(2):102-107. doi: 10.5830/CVJA-2020-052. Epub 2021 Jan 15. PMID 33496721
- [Result] AlTurki A, Essebag V. Atrial Fibrillation Burden: Impact on Stroke Risk and Beyond. Medicina (Kaunas). 2024 Mar 26;60(4):536. doi: 10.3390/medicina60040536. PMID 38674182
- See also: Groundbreaking consensus statement on conduction system pacing released: a major milestone in the evolution of pacing therapy — https://www.escardio.org/The-ESC/Press-Office/Press-releases/Groundbreaking-consensus-statement-on-conduction-system-pacing-released-a-major-milestone-in-the-evolution-of-pacing-therapy#